CLINICAL TRIAL: NCT01019317
Title: A Phase II Study of Twice Daily Cytarabine and Fludarabine in Acute Myelogenous Leukemia and High-Risk Myelodysplastic Syndrome
Brief Title: Fludarabine and Cytarabine in Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0781
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2013-10

CONDITIONS: Leukemia; AML; MDS; CML
Keywords: Acute Myelogenous Leukemia; High-Risk Myelodysplastic Syndrome; Chronic myeloid leukemia; CML; Blast crisis; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; Arabinosine Hydrochloride; Fludarabine; Fludarabine Phosphate; Fludara; Gemtuzumab Ozogamicin; Mylotarg
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — Cytarabine; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cytarabine + Fludarabine (Experimental): Fludarabine 15 mg/m^2 intravenous (IV) every 12 hours for 5 days; Cytarabine 0.5 grams/m^2 IV over 2 hours every 12 hours for 5 days.
  Interventions: Drug: Cytarabine; Drug: Fludarabine

INTERVENTIONS:
Drug: Cytarabine — 0.5 grams/m^2 over 2 hours(+/- 15 minutes) IV every 12 (+/-2) hours for 5 days (4 days in patients > 65 years and 3 days in patients with Eastern Cooperative Oncology Group (ECOG) performance status (PS) > 3).
  Other Names: Ara-C; Cytosar; DepCyt; Cytosine arabinosine hydrochloride
Drug: Fludarabine — 15 mg/m^2 to be given IV over 15-30 minutes every 12 (+/- 2) hours for 5 days. (4 days in patients > 65 years and 3 days in patients with PS > 3).
  Other Names: Fludara; Fludarabine Phosphate

SUMMARY:
The goal of this clinical research study is to learn if the combination of fludarabine and cytarabine can help to control Acute Myelogenous Leukemia (AML), High-Risk Myelodysplastic Syndrome (MDS) or Chronic Myeloid Leukemia (CML) in myeloid blast crisis. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs Fludarabine is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells). This may increase the likelihood of the cells dying.

Cytarabine is designed to insert itself into DNA and stop the DNA from repairing itself.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive fludarabine and cytarabine.

During each cycle (about 4-6 weeks), you will receive the study drugs for up to 5 days and you will be watched by the study staff for about 1 month.

Induction (Cycle 1):

For 3, 4, or 5 days during Days 1-5 of Cycle 1, you will receive fludarabine by vein over 15-30 minutes 2 times a day (about every 12 hours).

For 3, 4, or 5 days during Days 1-5 of Cycle 1, you will receive cytarabine by vein over about 2 hours 2 times a day (about every 12 hours).

If the cancer does not completely respond after Cycle 1, you may repeat induction (Cycle 1).

If the cancer completely responds, you will begin the consolidation cycles.

Consolidation (Cycles 2-7):

For 3 or 4 days during Days 1-4 of Cycles 2-7, you will receive fludarabine by vein over 15-30 minutes 2 times a day (about every 12 hours).

For 3 or 4 days during Days 1-4 of Cycles 2-7, you will receive cytarabine by vein over about 2 hours 2 times a day (about every 12 hours).

Study Visits:

At each study visit, you will be asked about any side effects you may be having and about any other drugs you may be taking.

During Induction Therapy (Cycle 1):

* Blood (about 2 tablespoons) will be drawn for routine tests every 3-7 days.
* About Day 28, you may have a bone marrow aspirate to check the status of the disease.

During Consolidation Therapy (Cycles 2-7):

* Blood (about 2 tablespoons) will be drawn for routine tests every 1-2 weeks.
* You will have a bone marrow aspirate every 2-3 cycles to check the status of the disease.

Length of Study:

You will be able to receive the study drugs for up to about 8 months. You will be taken off study treatment if you have intolerable side effects, if the disease gets worse, or if the study doctor thinks it is in your best interest.

Long-Term Follow-Up:

Every 3 months for 2 years after you are off study treatment, you will be called and asked how you are feeling, about any side effects you may be having, and about another other drugs you may be taking.

Supportive Care:

Please talk with your doctor about drugs that you can or cannot take while you are on study.

This is an investigational study. Cytarabine is FDA approved and commercially available as a frontline (first) treatment for AML. Fludarabine is FDA approved and commercially available for the treatment of CLL.

The combination of these 2 drugs to treat AML, MDS, or CML in myeloid blast crisis is investigational.

Up to 150 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an Internal Review Board (IRB)-approved informed consent document.
2. Age >/= 12 years.
3. Diagnosis of AML [other than acute promyelocytic leukemia (APL)] with refractory/relapsed disease. Patients with newly diagnosed AML will be eligible if not a candidate for intensive chemotherapy. Patients with high-risk (intermediate-2 or high by IPSS or >/=10% blasts) MDS will also be eligible. Patients with chronic myeloid leukemia (CML) in blast crisis will be eligible as well.
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= 3 at study entry.
5. Organ function as defined below (unless due to leukemia):

   i. Serum creatinine </= 3 mg/dL; ii. Total bilirubin </= 3 mg/dL; iii. Alanine aminotransferase (ALT)(Serum Glutamic Pyruvate Transaminase (SGPT)) </= 5 times upper limit of normal (ULN) or </= 10 times ULN if related to disease.
6. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days . Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.

Exclusion Criteria:

1. Pregnant or breastfeeding females.
2. Diagnosis of acute promyelocytic leukemia (M3).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/23/2009 through 10/25/2010. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 151 participants enrolled, four (4) participants were excluded from the trial before treatment.
Period: Overall Study
Arm/Group | Cytarabine + Fludarabine
Started | 151
Completed | 147
Not Completed | 4
Not completed — Not Eligible | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cytarabine + Fludarabine
Number analyzed (Participants) | 151
Age, Continuous [Median (Full Range); unit: years] | 63 [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 88
Region of Enrollment [Number; unit: participants]
  United States | 151

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Complete Response
Description: Complete Response (CR) was defined as: Neutrophil count ≥ 1.0 ×109/L, Platelet count ≥ 100 ×109/L, Bone marrow aspirate ≤5% blasts and No extramedullary leukemia. Response evaluation following Induction Therapy (Cycle 1) and every 2-3 cycles during Consolidation Therapy (Cycles 2 - 7) where Cycle is 4-6 weeks.
Time Frame: Minimally 6 weeks (Cycle 1) up to 1 year (7 cycles)
Population: Of participants enrolled, 147 participants received treatment and were evaluable.
Measure: Number; unit: Participants
Arm/Group | Cytarabine + Fludarabine
Number analyzed (Participants) | 147
Participants | 34

ADVERSE EVENTS:
Time Frame: Two years, ten months.
Description: Of the 151 participants registered, four did not recieve treatment and were excluded from adverse event reporting.
Arm/Group | Cytarabine + Fludarabine
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 100/147
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytarabine + Fludarabine (N=147)
Nausea (Gastrointestinal disorders) | 34 (34)
Vomiting (Gastrointestinal disorders) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 20 (20)
Mucositis (Gastrointestinal disorders) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 15 (15)
Elevated Liver Function (Hepatobiliary disorders) | 16 (16)
Infection (Infections and infestations) | 78 (78)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes